CLINICAL TRIAL: NCT02673151
Title: 68-Ga PSMA 11 PET/CT for Detection of Recurrent Prostate Cancer After Initial Therapy in Patients With Elevated PSA
Brief Title: 68Ga-PSMA PET/CT in Detecting Prostate Cancer Recurrence in Patients With Elevated PSA After Initial Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35932; NCI-2016-00094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0076 (Other: OnCore)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Prostate Adenocarcinoma; PSA Failure; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA-11 PET/CT (Experimental): Patients receive 68gallium-labeled prostate-specific membrane antigen-11 (68-Ga-PSMA-11). Participant will be injected IV with 3 to 7 millicurie (mCi) of 68Ga-PSMA-11. Beginning 50 to 100 minutes later, a low-dose computed tomography (CT) scan will be obtained from vertex to mid thighs; followed by a static positron emission tomography (PET) scan over the same .
  Interventions: Procedure: Computed Tomography (CT) scan; Drug: 68Ga-PSMA-11; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Procedure: Computed Tomography (CT) scan — PET/CT scan using 68gallium-labeled prostate-specific membrane antigen-11 (68-Ga-PSMA-11).
  Other Names: Computerized Axial Tomography (CAT); CAT scan; Computed Tomography (CT); Computerized Tomography (CT); CT Scan; tomography
Drug: 68Ga-PSMA-11 — 68gallium-labeled prostate-specific membrane antigen-11 (68-Ga-PSMA-11), administered by intravenous (IV) injection.
  Other Names: 68gallium-labeled prostate-specific membrane antigen-11 (68-Ga-PSMA-11); 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-HBED-CC-PSMA; HBED-CC-PSMA; DFKZ-11; Heidelberg compound
Procedure: Positron Emission Tomography (PET) — PET/CT scan using 68gallium-labeled prostate-specific membrane antigen-11 (68-Ga-PSMA-11).
  Other Names: Positron Emission Tomography scan (PET-scan); Proton magnetic resonance spectroscopic imaging

SUMMARY:
The purpose of this research study is to see if recurrent prostate cancer can be identified using a special procedure called a positron emission tomography (PET) scan. PET/CT is used to describe information regarding the function, as well as location and size of a tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate 68Ga-PSMA-11 PET/CT for detection of recurrent prostate cancer after initial therapy in patients with elevated PSA. PSMA refers to prostate-specific membrane antigen.

Eligible participants will undergo baseline assessments at enrollment. Study participants will receive 68Ga-PSMA-11 and undergo a PET/CT. Participants will be contacted at 24 to 72 hours following the scan in order to capture potential late occurring adverse events. Clinical follow up of participant at 3 to 12 months following the scan in order to analyze secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven prostate adenocarcinoma
* Rising prostate-specific antigen (PSA) after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy)

  * Post radical prostatectomy (RP) - American Urology Association (AUA) recommendation

    * PSA greater than 0.2 ng/mL measured 6 to 13 weeks after RP
    * Confirmatory persistent PSA greater than 0.2 ng/mL (total of two PSA measurements greater than 0.2 ng/mL)
  * Post-radiation therapy -American Society for Radiation Oncology (ASTRO)-Phoenix consensus definition

    * A rise of PSA measurement of 2 or more ng/mL over the nadir
* Karnofsky performance status of ≥ 50 (or Eastern Cooperative Oncology Group [ECOG] / World Health Organization [WHO] equivalent)
* Able to provide written consent

Exclusion Criteria:

* Investigational therapy for prostate cancer.
* Unable to lie flat, still or tolerate a positron emission tomograpy (PET) scan.
* Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2019-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baratto L, Song H, Duan H, Hatami N, Bagshaw HP, Buyyounouski M, Hancock S, Shah S, Srinivas S, Swift P, Moradi F, Davidzon G, Iagaru A. PSMA- and GRPR-Targeted PET: Results from 50 Patients with Biochemically Recurrent Prostate Cancer. J Nucl Med. 2021 Nov;62(11):1545-1549. doi: 10.2967/jnumed.120.259630. Epub 2021 Mar 5. PMID 33674398

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (68Ga-PSMA-11 PET/CT): Patients receive 68Ga-PSMA-11. Participant will be injected IV with 3 to 7 mCi of 68Ga PSMA 11 Beginning 50 to 100 minutes later, a low dose CT will be obtained from vertex to mid thighs; followed by a static PET emission scan over the same.
  * 68Ga-PSMA-11: Given IV
  * Computed Tomography: Undergo 68Ga-PSMA-11 PET/CT
  * Positron Emission Tomography: Undergo 68Ga-PSMA-11 PET/CT
Period: Overall Study
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT)
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT)
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 54
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Confirmation of Prostate Cancer Recurrence by 68Ga-PSMA-11 PET/CT
Description: Participants had suspected prostate cancer recurrence, and were evaluated with 68Ga-PSMA-11 PET/CT and by conventional methodologies, eg, histopathology/biopsy and/or conventional imaging. The outcome will be reported as the percentage of participants for whom the 68Ga-PSMA-11 PET/CT scan was positive (confirmed by conventional methodologies) or negative (not confirmed by conventional methodologies). The outcome is reported as the number of participants without dispersion. Up to 1 year was allowed for result by the conventional methodology.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT)
Number analyzed (Participants) | 61
Participants
  Tumor-positive by 68Ga-PSMA-11 PET/CT | 46
  Tumor-negative by 68Ga-PSMA-11 PET/CT | 15

2. Secondary Outcome: 68Ga-PSMA-11 PET/CT Sensitivity and Specificity
Description: 68Ga-PSMA-11 PET/CT sensitivity and specificity were assessed by comparing 68Ga-PSMA-11 PET/CT scan results with conventional imaging follow-up and/or histopathology/biopsy within the following 1 year. Sensitivity is a percentage that estimates, within a group of participants, the proportion within that group that truly has a disease or condition. Specificity is a percentage that estimates, within a group of participants, the proportion within that group that truly does not have the disease or condition. The outcome is reported as the point estimates for sensitivity and specificity, given as percentages representing agreement between the 68Ga-PSMA-11 PET/CT scan result and the conventional assessment, and the 95% CI. A higher point estimate represents better agreement between the methodologies.
Time Frame: up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage point estimate
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT)
Number analyzed (Participants) | 61
percentage point estimate
  Sensitivity | 100.0 [96.3 to 100.0]
  Specificity | 86.8 [81.8 to 90.9]

3. Secondary Outcome: 68Ga-PSMA-11 PET/CT Predictive Value by Region
Description: Positive predictive value (PPV) is the probability that participants with a positive screening test truly have the disease, and negative predictive value (NPV) is the probability that participants with a negative screening test truly do not have the disease. Predictive Value for 68Ga-PSMA-11 PET/CT was assessed by evaluating scans of the prostate, pelvic lymph nodes, paraaortic lymph nodes, mediastinal lymph nodes, bone, and lung. The outcome is reported as the probability as a percentage and the 95% CI.
Time Frame: up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage point estimate
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT)
Number analyzed (Participants) | 61
percentage point estimate
  Positive predictive value (PPV) | 76.4 [68.0 to 83.5]
  Negative predictive value (NPV) | 100.0 [98.2 to 100.0]

4. Secondary Outcome: Overall 68Ga-PSMA-11 PET/CT Scan Quality Stratified by PSA Level
Description: Scan quality was assessed by sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) determinations for the 68Ga-PSMA-11 PET/CT scans in participants stratified by prostate-specific antigen (PSA) level in ng/mL. Stratification levels were as follows.
  * 0.2 to < 0.5
  * 0.5 to < 1.0
  * 1.0 to < 2.0
  * 2.0 to < 5.0
  * ≥ 5.0, The outcome is expressed as the Sensitivity, Specificity, PPV, and NPV values observed for the PSA level strata, with 95% confidence interval.
Time Frame: up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage point estimate
Groups:
- Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 0.2 to < 0.5 ng/m?; Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 0.5 to < 1.0 ng/mL; Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 1.0 to < 2.0 ng/mL; Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 2.0 to < 5.0 ng/mL; Diagnostic (68Ga-PSMA-11 PET/CT) for PSA ≥ 5.0 ng/mL: Patients receive 68Ga-PSMA-11. Participant will be injected IV with 3 to 7 mCi of 68Ga PSMA 11 Beginning 50 to 100 minutes later, a low dose CT will be obtained from vertex to mid thighs; followed by a static PET emission scan over the same.
  * 68Ga-PSMA-11: Given IV
  * Computed Tomography: Undergo 68Ga-PSMA-11 PET/CT
  * Positron Emission Tomography: Undergo 68Ga-PSMA-11 PET/CT
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 0.2 to < 0.5 ng/m? | Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 0.5 to < 1.0 ng/mL | Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 1.0 to < 2.0 ng/mL | Diagnostic (68Ga-PSMA-11 PET/CT) for PSA 2.0 to < 5.0 ng/mL | Diagnostic (68Ga-PSMA-11 PET/CT) for PSA ≥ 5.0 ng/mL
Number analyzed (Participants) | 16 | 13 | 4 | 11 | 17
percentage point estimate
  Positive predictive value (PPV) | 31.3 [11.0 to 58.7] | 75 [50.9 to 91.3] | 100.0 [39.8 to 100.0] | 82.1 [63.1 to 93.9] | 84.7 [73.0 to 92.8]
  Negative predictive value (NPV) | 100.0 [96.9 to 100.0] | 100.0 [91.2 to 100.0] | NA [NA to NA] — Insufficient number of participants with events. | 100.0 [78.2 to 100.0] | 100.0 [86.8 to 100.0]
  Sensitivity | 100.0 [47.8 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [92.9 to 100.0]
  Specificity | 91.4 [85.1 to 95.6] | 88.9 [75.9 to 96.3] | NA [NA to NA] — Insufficient number of participants with events. | 75.0 [50.9 to 91.3] | 74.3 [56.7 to 87.5]

ADVERSE EVENTS:
Time Frame: 3 days (per protocol).
Arm/Group | Diagnostic (68Ga-PSMA-11 PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02673151/Prot_SAP_000.pdf